CLINICAL TRIAL: NCT02447068
Title: A Proof of Concept, Investigator Blinded Study to Evaluate the Efficacy and Safety of a Novel Combination of a Home Narrow Band Ultraviolet B (NBUVB) Lamp With an Occlusive Dressing in Adult Subjects With Mild to Moderate Psoriasis Vulgaris
Brief Title: Luma Light System Proof of Concept Study in Subjects With Mild to Moderate Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Illumicure Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: L-001
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Occlusive Dressings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Non-treatment Control (No Intervention): Control arm will not have any intervention
- Occlusive Dressing (Active Comparator): An off-the-shelf dressing occlusive dressing will be used as an active comparator.
  Interventions: Device: Occlusive Dressing
- Luma Light (Active Comparator): A NBUVB light will be used as an active comparator.
  Interventions: Device: Luma Light
- Luma Light System (Experimental): The experimental arm will be a combination of an occlusive dressing and NBUVB light.
  Interventions: Device: Luma Light System

INTERVENTIONS:
Device: Luma Light System — The Luma Light System combines a NBUVB light with an occlusive dressing.
  Arms: Luma Light System
Device: Luma Light — NBUVB light
  Arms: Luma Light
Device: Occlusive Dressing — Off-the-shelf occlusive dressing
  Arms: Occlusive Dressing

SUMMARY:
This is a proof of concept, investigator blinded study to evaluate the efficacy and safety of a novel combination of a home narrow band ultraviolet B (NBUVB) lamp with an occlusive dressing in adult subjects with mild to moderate psoriasis vulgaris. Four interpatient arms will be used to compare the efficacy of combination of NBUVB with an occlusive dressing to the light alone and to dressing alone and no treatment. Ten patients will be enrolled in this 6 weeks study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race, 18 to 65 (inclusive) years of age.
* Verbal and written informed consent obtained from the subject.
* Has a clinical diagnosis of mild to moderate psoriasis at the Screening and Baseline visits.
* Has an IGA score of 2 or 3.
* Target plaque assessment (TPA) score between 6-9 and a score of at least 2 for each of the 3 different psoriasis signs and symptoms (erythema, plaque elevation, and scaling)
* Has at least 4 plaques of at least 10 cm2 with TPA scores not differing from each other by a score of more than 1
* Is in good general health as determined by the Investigator based on the subject's medical history, vital signs and physical examination.
* Females of childbearing potential must have negative urine pregnancy test results.
* Females of childbearing potential agree to use acceptable methods of contraception from the screening visit continuously until 30 days after end of treatment.
* Subject agrees to use only the Sponsor provided cleanser and lotion during the study period.
* Subject is willing and able to return for all study visits.

Exclusion Criteria:

* Presence of psoriasis that was previously treated with prescription medications prior to the Screening visit and was non-responsive to treatment, as determined by the Investigator.
* Presence of any concurrent skin condition that could interfere with the evaluation of the study device, as determined by the Investigator.
* Female who is pregnant, nursing an infant, or planning a pregnancy during the study period.
* Treatment with any investigational drug or device within 30 days or 5 half-lives (whichever is longer) prior to the Baseline visit, or concurrent participation in another clinical trial with an investigational drug or device.
* History of melanoma.
* Subject has any medical, social or psychological conditions that, in the opinion of the Investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Target Plaque Assessment | 6 weeks
  Local efficacy will be evaluated with a 0-4 point scale for three signs and symptoms of psoriasis: erythema, plaque elevation, and scaling.
Local Skin Reactions | 6 weeks
  Tolerability will be evaluated through assessment of selected local signs and symptoms at the article-application site: Burning/stinging, pain and pruritus. Each sign or symptom will be graded at Baseline and each subsequent visit using a 0-3 scale (0 = none, 1 = mild, 2 = moderate, or 3 = severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Redwood Family Dermatology, Santa Rosa, California, United States